CLINICAL TRIAL: NCT01054443
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Investigate the Efficacy and Safety of S-888711 Tablets Administered Once-daily for 42 Days to Adult Subjects With Relapsed Persistent or Chronic Immune Thrombocytopenia With or Without Prior Splenectomy
Brief Title: A Study to Investigate the Efficacy and Safety of Lusutrombopag (S-888711) Tablets Administered to Adults With Immune Thrombocytopenia (ITP)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated before the planned sample size was enrolled because results indicated that a higher dose was necessary to elicit an efficacy effect.
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0913M0621
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Immune Thrombocytopenia (ITP)
Keywords: Blood Platelet Disorders; Immune Thrombocytopenia (ITP); Low Platelet Count; Thrombocytopaenia; S-888711; Splenectomy; Thrombopoiesis; Hematologic Disease; Auto-immune thrombocytopenic Purpura; Relapsed Persistent or Chronic ITP; Idiopathic Thrombocytopenic Purpura; Thrombotic Thrombocytopenic Purpura (TTP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Blood Platelet Disorders; Thrombocytopenia; Hematologic Diseases; Purpura, Thrombotic Thrombocytopenic | interventions — lusutrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo tablets orally once a day for 42 days.
  Interventions: Drug: Placebo
- Lusutrombopag 0.5 mg (Experimental): Participants received 0.5 mg lusutrombopag orally once a day for 42 days.
  Interventions: Drug: Lusutrombopag
- Lusutrombopag 0.75 mg (Experimental): Participants received 0.75 mg lusutrombopag orally once a day for 42 days.
  Interventions: Drug: Lusutrombopag
- Lusutrombopag 1.0 mg (Experimental): Participants received 1.0 mg lusutrombopag orally once a day for 42 days.
  Interventions: Drug: Lusutrombopag

INTERVENTIONS:
Drug: Placebo — Tablet
  Arms: Placebo
Drug: Lusutrombopag — Tablet
  Other Names: MULPLETA®; S-888711
  Arms: Lusutrombopag 0.5 mg; Lusutrombopag 0.75 mg; Lusutrombopag 1.0 mg

SUMMARY:
The primary objective of this study was to assess the efficacy of 3 dose levels of lusutrombopag (0.5 mg, 0.75 mg, and 1.0 mg) and placebo on platelet count.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated written informed consent
* Males and females ≥ 18 years of age
* All subjects must agree to use barrier contraception
* Diagnosis of ITP
* Subjects > 60 years must have had a diagnostic bone marrow aspiration
* Relapsed persistent or chronic ITP status, with or without prior splenectomy (exception: in Hungary only splenectomized subjects will be enrolled), after having failed at least 1 prior ITP therapy (excluding TPO agonists) and have a platelet count < 30,000/μL if not taking medications or < 50,000/μL despite concomitant steroids or other ITP therapies, such as danazol or immunosuppressive drugs
* Subjects receiving steroid therapy must be on a stable dose
* Prothrombin time (PT) and activated partial thromboplastin time (aPTT) within 20% of the upper limit of normal (ULN)
* Subjects receiving stable dosages of cyclosporine A, mycophenolate mofetil, azathioprine, or danazol are allowed. The dosages of all these medications must be stable for at least 4 weeks prior to Visit 1 (Day 1)

Exclusion Criteria:

* History of clinically important hemorrhagic clotting disorder
* Females who are pregnant, lactating, or taking oral contraceptives
* History of alcohol/drug abuse or dependence within 1 year
* Use of the following drugs or treatment prior to Visit 1 (Day 1):

  * Within 12 weeks - alemtuzumab, multi-drug systemic chemotherapy, stem cell therapy;
  * Within 8 weeks - rituximab
  * Within 2 weeks - platelet transfusions or plasmapheresis treatment
  * Within 4 weeks - use of anti-platelet or anti-coagulant drugs
  * Within 1 week - Rho(D) immune globulin or intravenous immunoglobulin
* History of clinically significant cardiovascular or thromboembolic disease within 26 weeks prior to Screening
* Splenectomy within 4 weeks prior to Screening
* Clinically significant laboratory abnormalities

  * Hemoglobin < 10.0 g/dL for men or women, not clearly related to ITP
  * Absolute neutrophil count < 1000/mm^3
  * Abnormal peripheral blood smear
  * Total bilirubin > 1.5 x upper limit of normal
  * Alanine aminotransferase (ALT) > 1.5 x upper limit of normal
  * Aspartate aminotransferase (AST) > 1.5 x upper limit of normal
  * Creatinine > 1.5 x upper limit of normal
  * Human immunodeficiency virus (HIV) positive
  * Hepatitis A immunoglobulin M antibody (IgM HAV) positive, hepatitis B surface antigen (HbsAg) or hepatitis C antibody (HCV) positive
  * Thyroid stimulating hormone (TSH) > 1.5 x upper limit of normal
  * Free thyroxine (T4) > 1.5 x upper limit of normal
* Exposure to previous thrombopoietin (TPO) mimetics/agonists (e.g., eltrombopag,romiplostim, E5501 [AKR-501] or LGD-4665) within 4 weeks prior to Screening
* Subjects unresponsive to previous TPO mimetics/agonists (e.g., eltrombopag, romiplostim, E5501 [AKR-501] or LGD-4665)
* Exposure to an investigative medication within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03-18 (Actual); Primary Completion 2010-11-24 (Actual); Study Completion 2010-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (18):
- United States (18):
  - Investigator, Anaheim, California
  - Investigator, Los Angeles, California
  - Investigator, Washington D.C., District of Columbia
  - Investigator, Boynton Beach, Florida
  - Investigator, Jacksonville, Florida
  - Investigator, Atlanta, Georgia
  - Investigator, Riverdale, Georgia
  - Investigator, Metairie, Louisiana
  - Investigator, Bethesda, Maryland
  - Investigator, Boston, Massachusetts
  - Investigator, Jefferson City, Missouri
  - Investigator, Kansas City, Missouri
  - Investigator, New Brunswick, New Jersey
  - Investigator, New York, New York
  - Investigator, Cleveland, Ohio
  - Investigator, San Antonio, Texas
  - Investigator, Salt Lake City, Utah
  - Investigator, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1:1:1 ratio to 1 of 4 treatment groups to receive lusutrombopag 0.5 mg, 0.75 mg, or 1.0 mg or placebo administered orally once daily for 42 days. Randomization was stratified according to Screening platelet count (< 30,000 cells/μL or ≥ 30,000 cells/μL to < 50,000 cells/μL).
Period: Overall Study
Arm/Group | Placebo | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (18.24) | 59.2 (24.60) | 55.0 (23.40) | 43.2 (15.39) | 54.7 (20.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 4 | 12
  Male | 2 | 1 | 4 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 4 | 5 | 4 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 5 | 5 | 5 | 19
  Black or African American | 1 | 0 | 0 | 0 | 1
Platelet Count at Screening [Count of Participants; unit: Participants]
  < 30,000 cells /μL | 5 | 5 | 4 | 5 | 19
  ≥ 30,000 cells/μL to < 50,000 cells/μL | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Response
Description: Responders were participants with one of the following:
  1. achieved a platelet count of ≥ 50,000 cells/µL after 6 weeks of dosing; or
  2. prematurely withdrawn due to a platelet count > 400,000 cells/µL prior to Day 42.
  Participants were counted as non-responders if any of the following conditions held:
  * The above conditions were not satisfied;
  * They received rescue medications;
  * They satisfied the above conditions after receiving restricted medications during the treatment period;
  * They had achieved a platelet count of ≥ 50,000 cells/µL before Week 6 but not after Week 6; or
  * They withdrew for any reason other than a platelet count > 400,000 cells/µL.
Time Frame: Week 6
Population: The full analysis set included all randomized participants who received at least 1 dose of study drug and had a platelet count at Baseline and at least 1 platelet count after randomized study drug was taken.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
Number analyzed (Participants) | 5 | 5 | 5 | 5
percentage of participants | 0.0 [NA to NA] — Could not be estimated when number of responses = 0 | 20.0 [0.5 to 71.6] | 0.0 [NA to NA] — Could not be estimated when number of responses = 0 | 0.0 [NA to NA] — Could not be estimated when number of responses = 0
Statistical Analysis 1: Comparison: Placebo vs Lusutrombopag 0.5 mg vs Lusutrombopag 0.75 mg vs Lusutrombopag 1.0 mg; The primary efficacy evaluation was to test if there was a linear relationship existing such that the higher the dose level, the larger the percentage of responders. The Cochran-Armitage trend test was employed by assigning the score 0, 0.5, 0.75, and 1 to placebo, lusutrombopag 0.5, 0.75, and 1.0 mg group, respectively, at the 0.025 level of significance (1-sided) to determine the test statistic for detecting a dose-response in the percentage of responders; Test type: Other; p = 0.431, Cochran-Armitage Trend Test; Cochran-Armitage Trend Test Statistic = 0.173

2. Secondary Outcome: Change From Baseline in Platelet Count at Week 6
Time Frame: Baseline and Week 6
Population: Full analysis set participants who completed 6 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: cells/µL
Arm/Group | Placebo | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
Number analyzed (Participants) | 5 | 5 | 5 | 4
cells/µL | -3566.0 (6400.05) | 21978.1 (6095.54) | 8235.4 (6465.37) | -2809.4 (6866.08)
Statistical Analysis 1: Comparison: Placebo vs Lusutrombopag 0.5 mg; Test type: Other; LS Mean Difference = 25544.0, 95% CI 2-sided [6202.8 to 44885.3] — The difference of least squares means (LSMeans) between each of the lusutrombopag treatment groups and placebo was estimated after adjusting for the Baseline platelet count using analysis of covariance (ANCOVA)
Statistical Analysis 2: Comparison: Placebo vs Lusutrombopag 0.75 mg; Test type: Other; LS Mean Difference = 11801.3, 95% CI 2-sided [-8809.3 to 32411.9] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Lusutrombopag 1.0 mg; Test type: Other; LS Mean Difference = 756.6, 95% CI 2-sided [-18794.3 to 20307.5] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the percentage of the cumulative time a platelet count was ≥ 50,000 cells/µL during the treatment period.
Time Frame: 6 weeks
Population: Participants in the full analysis set with platelet counts ≥ 50,000 cells/μL at any time during the 6-week treatment period.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
Number analyzed (Participants) | 0 | 4 | 3 | 1
percentage of days |  | 0.399 [0.06 to 0.81] | 0.426 [0.33 to 0.55] | 0.103 [0.103 to 0.103]

4. Secondary Outcome: Percentage of Participants Who Achieved a Platelet Count of ≥ 30,000 Cells/µL and Doubled the Baseline Platelet Count After 6 Weeks of Dosing
Time Frame: Week 6
Population: Participants in the full analysis set who completed 6 weeks of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
Number analyzed (Participants) | 5 | 5 | 5 | 4
percentage of participants | 0.0 | 60.0 | 20.0 | 0.0

5. Secondary Outcome: Percentage of Participants Who Achieved a Platelet Count of ≥ 50,000 Cells/µL and Doubled the Baseline Platelet Count After 6 Weeks of Dosing
Time Frame: Week 6
Population: Participants in the full analysis set who completed 6 weeks of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
Number analyzed (Participants) | 5 | 5 | 5 | 4
percentage of participants | 0.0 | 40.0 | 0.0 | 0.0

6. Secondary Outcome: Number of Participants With Worst Severity of Bleeding Associated With ITP During the Treatment Period,
Description: Bleeding assessments were performed by the Investigator according to the World Health Organization (WHO) criteria bleeding scale:
  Grade 0: no bleeding; Grade 1: petechial bleeding; Grade 2: mild blood loss (clinically significant); Grade 3: gross blood loss, requires transfusion (severe); Grade 4: debilitating blood loss, retinal or cerebral associated with fatality.
  For each participant, the most severe WHO bleeding grade observed during the 6-week treatment period is reported.
Time Frame: 6 weeks
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants
  Grade 0 | 0 | 0 | 2 | 0
  Grade 1 | 2 | 3 | 2 | 3
  Grade 2 | 3 | 2 | 1 | 2
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Who Received Rescue Medication During the Treatment Period
Time Frame: 6 weeks
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 1 | 2 | 3 | 2

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a subject administered a pharmaceutical product during the course of a clinical investigation, including any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product (IP), whether or not thought to be related to the IP. AEs reported after initial study drug administration were considered treatment-emergent.
  A serious adverse event is defined as any AE that resulted in death, was life-threatening, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect or an important medical event that, based upon medical judgment, may jeopardize the participant or require medical or surgical intervention to prevent one of the outcomes listed above.
  A treatment-related AE is any AE determined by the investigator to be possibly related, probably related, or definitely related to study drug.
Time Frame: 6 weeks
Population: The safety population included all participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants
  Any treatment-emergent adverse event | 4 | 5 | 5 | 4
  Serious adverse events | 0 | 0 | 0 | 1
  Treatment-related adverse events | 1 | 1 | 0 | 2
  Treatment-related serious adverse events | 0 | 0 | 0 | 0
  Adverse events leading to withdrawal of study drug | 0 | 0 | 0 | 0

9. Secondary Outcome: Lusutrombopag Plasma Concentration
Description: Plasma concentrations of lusutrombopag were determined using a validated liquid chromatography mass spectrometry method. The lower limit of quantification (LOQ) for the plasma assay for lusutrombopag was 0.1 ng/mL.
Time Frame: Days 8, 22, and 36, after dosing
Population: Participants who received at least 1 dose of study drug
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
Number analyzed (Participants) | 5 | 5 | 5
ng/mL
  Day 8: number analyzed (Participants) | 5 | 5 | 4
  Day 8 | 16.5 (35.40) | 21.7 (52.77) | 33.3 (32.74)
  Day 22: number analyzed (Participants) | 5 | 5 | 3
  Day 22 | 19.1 (32.10) | 19.6 (32.20) | 30.7 (42.97)
  Day 36: number analyzed (Participants) | 5 | 5 | 4
  Day 36 | 24.1 (14.22) | 21.1 (36.33) | 30.4 (40.28)

10. Secondary Outcome: Plasma Concentration of Metabolite S-888711 Deshexyl
Description: Plasma concentrations of the major metabolite S-888711 deshexyl were determined using a validated liquid chromatography mass spectrometry method. The lower limit of quantification (LOQ) for the plasma assay for S-888711 deshexyl was 0.1 ng/mL.
Time Frame: Days 8, 22, and 36, after dosing
Population: Participants who received at least 1 dose of study drug, with available data at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
Number analyzed (Participants) | 5 | 5 | 5
ng/mL
  Day 8: number analyzed (Participants) | 4 | 5 | 4
  Day 8 | 0.1 (68.10) | 0.3 (176.69) | 0.2 (50.41)
  Day 22: number analyzed (Participants) | 5 | 5 | 3
  Day 22 | 0.1 (23.87) | 0.2 (141.38) | 0.2 (50.20)
  Day 36: number analyzed (Participants) | 5 | 5 | 4
  Day 36 | 0.1 (28.15) | 0.2 (154.49) | 0.2 (101.93)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Placebo | Lusutrombopag 0.5 mg | Lusutrombopag 0.75 mg | Lusutrombopag 1.0 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 1/5
Other Adverse Events (participants affected / at risk) | 4/5 | 5/5 | 5/5 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Lusutrombopag 0.5 mg (N=5) | Lusutrombopag 0.75 mg (N=5) | Lusutrombopag 1.0 mg (N=5)
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Lusutrombopag 0.5 mg (N=5) | Lusutrombopag 0.75 mg (N=5) | Lusutrombopag 1.0 mg (N=5)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Cyst (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Muscle spasms (General disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Clumsiness (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Victim of sexual abuse (Social circumstances) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.